CLINICAL TRIAL: NCT01154790
Title: A Randomized, Double-blind Study Evaluating the Upper Gastrointestinal Safety on Multiple Doses of CG100649 in Healthy Subjects
Brief Title: Phase I Study on Multiple Oral Dosing of CG100649
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CG100649-1-04
Record Dates: First submitted 2010-06-16; First posted 2010-07-01 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — CG100649; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CG100649 (Experimental): By the amount of doses, the groups are classified
  Interventions: Drug: CG100649; Drug: Placebo
- Naproxen (Active Comparator): By the amount of doses, the groups are classified
  Interventions: Drug: Placebo; Drug: Naproxen
- Placebo (Placebo Comparator): By the amount of doses, the groups are classified
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CG100649 — 6 subjects: study drug 2 subjects: placebo
  Arms: CG100649
Drug: Placebo — 6 subjects: study drug 2 subjects: placebo
Drug: Naproxen — 6 subjects: study drug 2 subjects: placebo
  Other Names: NAXEN
  Arms: Naproxen

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and pharmacokinetics of 3 escalating loading and maintenance dose regimens of CG100649 administered orally for 7 total days in healthy volunteers.

DETAILED DESCRIPTION:
Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information if used CTCAE and normal ranges if relevant.

ELIGIBILITY:
Inclusion Criteria:

1. 19-55 years old. Body weight is over 50 kg (male) and over 45 kg (female). Body weights must be within 20% of ideal body weight for their height according to the ideal body weight table.
2. No significant congenital/chronic disease. No symptoms in physical examination.
3. Appropriate subjects as determined by past medical history, laboratory tests, serology and urinalysis.
4. Be able to understand the objective, method of the study, the characteristics of investigational drug, and comply with the requirement of the study. Subject must provide written informed consent prior to study participation.

Exclusion Criteria:

1. History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or cognitive disorders.
2. History of gastrointestinal disorders (bleeding, ulceration, hemorrhoids, piles) or disorders of absorption, distribution, metabolism, excretion.
3. History of known hypersensitivity to drugs including CG100649.
4. After taking a rest in sitting position for 3 minutes, subjects who have low blood pressure (Systolic BP ≤ 90 mmHg or Diastolic BP ≤ 50 mmHg) or high blood pressure (Systolic BP ≥ 150 mmHg or Diastolic BP ≥ 100 mmHg).

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety (normal results for safety tests) | 27days
  Cardiovascular: BP,ECG, Holter monitoring
  GI: Fecal occult blood
  Kidney: Urine electrolyte test
  Adverse events
  Physical examination, vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Seonggu Ro, Study Director — CrystalGenomics, Inc.
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided